CLINICAL TRIAL: NCT07286292
Title: A Phase 2, Single Arm, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Vorasidenib in Pediatric Participants Aged 12 to < 18 Years Old With Grade 2 Astrocytoma or Oligodendroglioma With an IDH1 or IDH2 Mutation
Brief Title: Vorasidenib Study in Pediatric Participants With Grade 2 Astrocytoma or Oligodendroglioma With an IDH1 or IDH2 Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (I.R.I.S.) (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S095032-236
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Grade 2 Astrocytoma or Oligodendroglioma With an IDH1 or IDH2 Mutation
MeSH Terms: interventions — vorasidenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Vorasidenib (Experimental)
  Interventions: Drug: Vorasidenib

INTERVENTIONS:
Drug: Vorasidenib — 40mg taken orally daily for participants weighing ≥ 40 kg OR 20mg taken orally daily for participants weighing ≥ 25 kg to < 40 kg

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, efficacy profile, and effect on growth and development of vorasidenib in pediatric participants aged 12 to < 18 years old with grade 2 glioma with an IDH1 or IDH2 mutation. The study includes a screening period, a treatment period consisting of continuous 28-day cycles of treatment, a safety follow-up period and a long-term follow-up period. The long-term follow-up period will assess participants for growth, development, and long-term safety impacts for approximately 5 years after the start of treatment or until Tanner Stage V is reached (whichever is later). Participants may undergo blood tests, heart tests (electrocardiogram (ECG)), imaging (MRI, X-ray), vital sign checks, and physical exams.

ELIGIBILITY:
Inclusion Criteria:

* Weigh ≥ 25 kg at Screening.
* Written informed consent/assent must be obtained from a legally authorized representative, and assent must be obtained from the participant in accordance with local regulations. Participants and their families must be willing and able to comply with the scheduled visits, treatment plans, procedures, and laboratory tests, including serial peripheral blood sampling, during the study.
* Have Grade 2 astrocytoma or oligodendroglioma per World Health Organisation (WHO) 2021 criteria.
* Have had at least 1 prior surgery for glioma (biopsy, sub-total resection, gross-total resection) and no other prior anticancer therapy, including chemotherapy and radiotherapy, and do not need immediate chemotherapy or radiotherapy in the opinion of the Investigator.
* Have:
* Confirmed IDH1 or IDH2 gene mutation, as well as known 1p19q and/or ATRX (Alpha Thalassemia/Mental Retardation Syndrome X-linked) status based on local testing of tumor tissue by an accredited laboratory.
* For astrocytoma: Absence of 1p19q co-deletion and/or documented loss of nuclear ATRX expression or ATRX mutation by local testing.
* For oligodendroglioma: Presence of 1p19q co-deletion by local testing.
* Have magnetic resonance imaging (MRI)-evaluable, measurable, non-enhancing disease
* Have a Karnofsky Performance Score (KPS; for participants ≥ 16 years of age) or Lansky Play-Performance Scale (LPPS; for participants < 16 years of age) score of ≥ 70. Karnofsky Performance Score and LPPS < 70 due to functional limitations as a result of prior surgical resections or due to the anatomical location of the tumor will be permitted.
* Have adequate bone marrow function as evidenced by:
* Absolute neutrophil count ≥ 1500/mm3 or ≥ 1.5 × 109/L
* Hemoglobin ≥ 9 g/dL
* Platelets ≥ 100,000/mm3 or ≥ 100 × 109/L
* Have adequate hepatic function as evidenced by:
* Serum total bilirubin ≤ 1.5 × ULN; if > 1.5 ULN and due to Gilbert syndrome, total bilirubin ≤ 3 × ULN with direct bilirubin ≤ ULN
* AST at or below ULN and ALT at or below ULN
* Alkaline phosphatase (ALP) ≤ 2.5 × ULN
* Have adequate renal function as evidenced by:
* Serum creatinine ≤ 2.5 × ULN, OR
* eGFR > 40 mL/min/1.73 m2 based on the Bedside Schwartz method 0.413 × (Height in cm/Serum Creatinine in mg/dL)
* Have recovered from any clinically relevant toxicities associated with any prior surgery for the treatment of glioma unless stabilized under medical management (functional limitations as a result of prior surgical resections or due to the anatomical location of the tumor will be permitted).
* Female participants of reproductive potential must have a negative serum pregnancy test before starting investigational medicinal product (IMP).
* Women of childbearing potential as well as fertile male participants with female partners of reproductive potential, must agree to abstain from sexual intercourse or to use 2 effective methods of contraception from screening until at least 90 days after the last dose of IMP.

Exclusion Criteria:

* Have had any prior anticancer therapy other than surgery (biopsy, sub-total resection, gross-total resection) for treatment of glioma including, but not limited to, systemic chemotherapy, radiotherapy, vaccines, small molecule inhibitors, IDH inhibitors, and investigational agents.
* Have features assessed as high-risk by the Investigator.
* Have leptomeningeal disease.
* Concurrent active malignancy except for curatively resected nonmelanoma skin cancer or curatively treated carcinoma in situ. Participants with previously treated malignancies are eligible provided they have been disease-free for 3 years at Screening.
* Unable to swallow oral medication.
* Are pregnant or breastfeeding.
* Are participating in another interventional study at the same time; participation in non-interventional registries or epidemiological studies is allowed.
* Have a severe or uncontrolled active acute or chronic infection or an unexplained fever > 38.5°C within 7 days of C1D1.
* Have a known hypersensitivity to any of the components of vorasidenib.
* Have significant active cardiac disease within 6 months before the start of IMP, including New York Heart Association Class III or IV congestive heart failure, myocardial infarction, unstable angina, and/or stroke.
* Have a heart-rate corrected QT interval using Fridericia's formula (QTcF) ≥ 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events.
* Are taking therapeutic doses of steroids (defined as > 1.5 mg/day dexamethasone or >10 mg/day prednisone or equivalent) for signs/symptoms of glioma. Participants taking physiologic doses (defined as ≤ 1.5 mg/day dexamethasone or ≤ 10 mg/day prednisone or equivalent) for medical conditions not related to glioma will be permitted.
* Are taking any medications that are CYP2C19 or CYP3A substrates with a narrow therapeutic index or strong inhibitors of CYP1A2.
* Have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, known positive human immunodeficiency virus (HIV) antibody results, or AIDS-related illness. Participants with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Participants with chronic HBV or HIV that is adequately suppressed by institutional practice will be permitted.
* Have known active inflammatory gastrointestinal disease, chronic diarrhea, previous gastric resection or lap band dysphagia, short-gut syndrome, gastroparesis, or other condition that limits the ingestion or gastrointestinal absorption of drugs administered orally. Gastroesophageal reflux disease under medical treatment is allowed (assuming no drug interaction potential).
* Have any other acute or chronic medical or psychiatric condition.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2033-05-02 (Estimated); Study Completion 2033-05-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events (AEs) leading to discontinuation, or Adverse Events (AEs) leading to death | From start of treatment through 28 days after last dose for AEs (Safety follow-up), study-related SAEs will be reported through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Severity of AEs | From start of treatment through 28 days after last dose for AEs (Safety follow-up), study-related SAEs will be reported through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
  As assessed by the NCI-CTCAE version 5.0.
Height and Weight Percentiles at Study Visits | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Change in Height and Weight Percentiles from Cycle 1 Day 1 (C1D1) | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Tanner staging | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
  Tanner stages represent puberty progression from stage 1 being the prepubertal form to stage 5 representing the final adult form.
Average age of menarche | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
  Historically and/or while on treatment, if applicable
Change from C1D1 to the worst on-treatment value of leutenizing hormone (LH) | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Change from C1D1 to the worst on-treatment value of follicle-stimulating hormone (FSH) | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Change from C1D1 to the worst on-treatment value of anti-Müllerian hormone (AMH) | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Change from C1D1 to the worst on-treatment value of estradiol | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
  For females only
Change from C1D1 to the worst on-treatment value of testosterone | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
  For males only
Change from C1D1 to the worst on-treatment value of Insulin-like growth factor 1 (IGF-1) | Cycle 1 Day 1 (C1D1) (each cycle is 28 days long)
Change from C1D1 to the worst on-treatment value of Insulin-Like Growth Factor-Binding Protein 3 (IGFBP-3) | Cycle 1 Day 1 (C1D1) (each cycle is 28 days long)
Change from C1D1 to the worst on-treatment value of thyroid stimulating hormone (TSH) | Cycle 1 Day 1 (C1D1) (each cycle is 28 days long)
Change from C1D1 to the worst on-treatment value of Free T4 (thyroxine) | Cycle 1 Day 1 (C1D1) (each cycle is 28 days long)
Change from C1D1 to the worst on-treatment hand/wrist bone age as determined by X-ray | From start of treatment through long-term follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through PFS follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Objective response (OR) | Through PFS follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Best overall response of complete response (CR), partial response (PR), or minor response (mR) | Through PFS follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Time to response (TTR) | Through PFS follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Time to CR, PR, or mR | Through PFS follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Duration of response (DoR) | Through PFS follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Duration of CR, PR, or mR | Through PFS follow-up (approximately 5 years per participant for a total study duration of approximately 7 years)
Plasma concentration of vorasidenib | Through Cycle 3 Day 1 (C3D1) (each cycle is 28 days long)
Plasma concentration of AGI-69460 | Through Cycle 3 Day 1 (C3D1) (each cycle is 28 days long)

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.